CLINICAL TRIAL: NCT06293534
Title: Thyroid Dysfunction in Patient With Major Psychiatric Disorders Admitted to Psychiatric Unit of Assiut University Hospital
Brief Title: Thyroid Dysfunction in Patients With Major Psychiatric Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Mahmoud Abdelsalam, Principle Investigator, Assiut University
Other Study IDs: PsychThyroid
Record Dates: First submitted 2023-12-13; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Thyroid Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with major psychiatric disorders: Patients diagnosed with major psychiatric disorders according to the Diagnostic Statistical Manual version 5 (DSM 5-TR), admitted to the psychiatry department in Assiut University Hospital.
  Interventions: Diagnostic Test: TSH,T3,T4

INTERVENTIONS:
Diagnostic Test: TSH,T3,T4 — Diagnosis of the psychiatric disorders among study group will be assessed and recorded and history of Electroconvulsive therapy (ECT) also will be recorded , physical examination for signs that suggests actual thyroid disease such as unexplained bradycardia or tachycardia, hypothermia , goiter or non palpable thyroid among study group will be assessed

SUMMARY:
Thyroid dysfunction in major psychiatric disorders in psychiatric patients admitted to psychiatric unit of assiut university hospital

DETAILED DESCRIPTION:
Thyroid hormones play a key role in the development, metabolism and functioning of many organs and have a profound influence on the human brain and behaviour. the coexistence of thyroid insufficiency with mental disorders was recognized . Mental disorders accounted for 6 of the 20 leading causes of disability worldwide for the most productive section of the population.Thyroid diseases can present with various neuropsychiatric manifestations which include mood, anxiety, psychotic, and cognitive disorders.Thus, thyroid function tests are routinely checked in psychiatric patients, While dealing with neurocognitive or neuropsychiatric manifestations,thyroid disorders should be ruled out by appropriate thyroid function tests which include Thyroid-stimulating hormone (TSH), free T3, free T4 and reverse T3.Multiple studies on the prevalence of thyroid dysfunctions on psychiatric patients in different populations were done and reported .the presence of thyroid dysfunction in patients with schizophrenia-spectrum disorder as well as mood disorders .Mental disorders merge highly with thyroid disease.Bio-psycho-social medical model are important for treatment of mental disorders associated with thyroid dysfunction .Till now, there is no literature on the rates of thyroid dysfunction among psychiatric patient in our population in assiut university hospital which can be helpful in the proper management of the cases.

ELIGIBILITY:
Inclusion Criteria:

* patients with major psychiatric disorders admitted to psychiatric unit of neuropsychiatry department of Assiut university hospital in Egypt.

Exclusion Criteria:

* pregnant or lactating females
* Patients on estrogen therapy or contraceptive
* Patients on carbamazepine, oxcarbazepine, phenytoin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mental illness, diagnosed based on DSM 5-TR and whose condition is severe enough to require admission in the psychiatric ward.
Sampling Method: Probability Sample
Enrollment: 173 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
the level of thyroid hormones among psychiatric patients | One year
  TSH, free T3 and free T4 levels in psychiatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Abdelrahman mohamed, M.D., Study Director — Assiut University; Rania Mohamed Mahmoud Hafez, M.D., Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kamble MT, Nandedkar PD, Dharme PV, L LS, Bhosale PG. Thyroid function and mental disorders: an insight into the complex interaction. J Clin Diagn Res. 2013 Jan;7(1):11-4. doi: 10.7860/JCDR/2012/4861.2656. Epub 2013 Jan 1. PMID 23449617
- [Background] Lekurwale V, Acharya S, Shukla S, Kumar S. Neuropsychiatric Manifestations of Thyroid Diseases. Cureus. 2023 Jan 20;15(1):e33987. doi: 10.7759/cureus.33987. eCollection 2023 Jan. PMID 36811059
- [Background] Dickerman AL, Barnhill JW. Abnormal thyroid function tests in psychiatric patients: a red herring? Am J Psychiatry. 2012 Feb;169(2):127-33. doi: 10.1176/appi.ajp.2011.11040631. PMID 22318794
- [Background] Lederbogen F, Hermann D, Hewer W, Henn FA. Thyroid function test abnormalities in newly admitted psychiatric patients residing in an iodine-deficient area: patterns and clinical significance. Acta Psychiatr Scand. 2001 Oct;104(4):305-10. doi: 10.1034/j.1600-0447.2001.00328.x. PMID 11722306
- [Background] Radhakrishnan R, Calvin S, Singh JK, Thomas B, Srinivasan K. Thyroid dysfunction in major psychiatric disorders in a hospital based sample. Indian J Med Res. 2013 Dec;138(6):888-93. PMID 24521631
- [Background] Fukao A, Takamatsu J, Arishima T, Tanaka M, Kawai T, Okamoto Y, Miyauchi A, Imagawa A. Graves' disease and mental disorders. J Clin Transl Endocrinol. 2019 Oct 11;19:100207. doi: 10.1016/j.jcte.2019.100207. eCollection 2020 Mar. PMID 31763175